CLINICAL TRIAL: NCT01046266
Title: An Exploratory, Open Label Multicenter Study to Investigate Pharmacodynamic of RO5083945, a Human Monoclonal Antibody Antagonist of Epidermal Growth Factor Receptor (EGFR), Compared to Cetuximab in Patients With Operable Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Pharmacodynamics of RO5083945 in Patients With Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22350; 2009-012656-25
Record Dates: First submitted 2009-11-16; First posted 2010-01-11 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — imgatuzumab; Cetuximab

ARMS (2):
- A (Experimental)
  Interventions: Drug: RO5083945
- B (Active Comparator)
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: RO5083945 — 700mg iv weekly
  Arms: A
Drug: cetuximab — 400mg/m2 iv 1st dose, 250mg/m2 iv subsequent weekly doses
  Arms: B

SUMMARY:
This open-label study will assess the pharmacodynamics, safety and efficacy of RO5083945 as compared to cetuximab in patients with head and neck squamous cell carcinoma. Patients will receive at least 2 infusions of either RO5083945 or cetuximab. Anticipated time on study treatment is up to 3 months, and target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx

Exclusion Criteria:

* carcinoma of nasal cavity, paranasal sinus and nasopharynx
* recurrent squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx
* known positivity for HIV, hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
immune cell infiltration head and neck squamous cell cancer (HNSCC) | through study completion or early study discontinuation

SECONDARY OUTCOMES:
pharmacodynamics: T lymphocytes, B lymphocytes, NK cells, plasma cytokine levels | through study completion or early study discontinuation
safety and efficacy: AEs, laboratory parameters, tumour assessments | through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- France (2):
  - Toulouse
  - Villejuif
- Milan, Lombardy, Italy
- Nijmegen, Netherlands
- Spain (2):
  - Barcelona, Barcelona
  - Seville, Sevilla
- London, United Kingdom

REFERENCES:
- [Derived] Temam S, Spicer J, Farzaneh F, Soria JC, Oppenheim D, McGurk M, Hollebecque A, Sarini J, Hussain K, Soehrman Brossard S, Manenti L, Evers S, Delmar P, Di Scala L, Mancao C, Feuerhake F, Andries L, Ott MG, Passioukov A, Delord JP. An exploratory, open-label, randomized, multicenter study to investigate the pharmacodynamics of a glycoengineered antibody (imgatuzumab) and cetuximab in patients with operable head and neck squamous cell carcinoma. Ann Oncol. 2017 Nov 1;28(11):2827-2835. doi: 10.1093/annonc/mdx489. PMID 28950289